CLINICAL TRIAL: NCT03575442
Title: "Art Therapy" in Acute Psychiatry: a Psychosocial Intervention
Brief Title: "Art Therapy" in Acute Psychiatry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CHUC-007-17
Record Dates: First submitted 2018-05-24; First posted 2018-07-02 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia; Mood Disorders; Mental Disorder; Nurse-Patient Relations
MeSH Terms: conditions — Schizophrenia; Mood Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3 session program of "art therapy" (Other): Development of the program applied as a group, during three weeks, one session a week, each lasting approximately 90 minutes and assisted by a specialist in plastic expression. Each session was held in an occupational therapy room, including all the material deemed necessary for the execution of some of the techniques introduced by the technician. After each session, a semi-structured interview was conducted with each participant in order to analyze the meanings attributed.
  Interventions: Behavioral: 3 session program of "art therapy"

INTERVENTIONS:
Behavioral: 3 session program of "art therapy" — With this program, we expect to offer socio-emotional well-being in the psychiatric context, and creative self-expression through painting. In addition, we hope to provide contributions towards the creation of quality standards of the professional practice of nurses, within the context of implementing psychosocial programs in mental health.

SUMMARY:
Background: Given the complexity of this problem, psychiatric in-patients in the acute stage of their disease need different types of therapeutic programs to recover they mental health state. Usually they're submitted to systematic biological programs (namely psychopharmaceuticals), often considered a priority when compared to psychosocial programs. Among the different therapies that have been introduced in this context "art therapy", also named creative therapy, can constitute a treatment that complements the allopathic treatments, providing improvements in self-esteem and self-efficiency, distraction and relief from concerns and negative thoughts. Scientific evidence on the effects of psychosocial programs in the context of hospitalization of acute cases is scarce.

Aims: a) evaluate the effectiveness of a 3 session program of "art therapy" in changing emotional indicators, namely depression, anxiety, stress, and psychological well-being, in individuals with mental illness; b) analyze the meanings a person attributes to his creative self-expression.

Method: This is a pre-experimental, prospective study, with a pre test-post test design without control group, with a mixed approach (quantitative and qualitative). The study was performed in the psychiatry unit (Psiquiatria B), in the Centro Hospitalar e Universitário de Coimbra - Portugal. The target population was composed by men (older than 18), hospitalized in this ward. The exclusion criteria were: individuals with active psychotic symptomology, in manic phase and/or refusing to participate. The instruments used to collect information were: Depression, Anxiety and Stress Scale [DASS-21]; Ryff Scales of Psychological Well-Being (SPWB - 18 item version) and a semi-structured interview.

Data collection and the development of this study occurred in the following manner:

* Initial evaluation to verify the sample selection criteria in the first 48 hours after patient hospitalization;
* Obtain informed consent for the application of instruments and participation in the "art therapy" intervention program;
* Application of instruments (DASS-21 and SPWB-18 item version) before intervention;
* Development of the program applied as a group, during three weeks, one session a week, each lasting approximately 90 minutes and assisted by a specialist in plastic expression. Each session was held in an occupational therapy room, including all the material deemed necessary for the execution of some of the techniques introduced by the technician. After each session, a semi-structured interview was conducted with each participant in order to analyze the meanings attributed.
* In the end of the program, the same instruments were reapplied.

ELIGIBILITY:
Inclusion Criteria:

* men (older than 18), hospitalized in a psychiatric unit;
* capable of communicating and understanding communication;
* acceptance and commitment to participate in the study;
* signature of study informed consent.

Exclusion Criteria:

* individuals with active psychotic symptomology, in manic phase and/or refusing to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the participant's emotional states of depression, anxiety and stress | Post-intervention assessment (week 3)
  Outcome measure - Depression, Anxiety and Stress Scale [DASS-21] - (Lovibond et al.,1995 adapted by Apóstolo, Mendes & Azeredo, 2006)
Change from Baseline in the participant's psychological well-being | Post-intervention assessment (week 3)
  Outcome measure - Ryff Scales of Psychological Well-Being (SPWB - 18 item version) - (Ryff, 1989 adapted by Novo, Neto, Marcelino & Santo, 2006)
Semi-structured interview | Post-intervention assessment (week 3)
  Aim: explore in a psychiatric context [in the acute stage of the disease] the sick person's experiences related to expression by painting after each of three scheduled interviews, during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Clara A. Campos, RN, Principal Investigator — Unidade Local de Saúde de Coimbra, EPE
Locations (1):
- Psiquiatria B - Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

REFERENCES:
- [Background] Stickley T, Hui A. Arts In-Reach: taking 'bricks off shoulders' in adult mental health inpatient care. J Psychiatr Ment Health Nurs. 2012 Jun;19(5):402-9. doi: 10.1111/j.1365-2850.2011.01811.x. Epub 2011 Sep 20. PMID 22070164
- [Background] Van Lith, T. Art therapy in mental health: A systematic review of approaches and practices. The Arts in Psychotherapy. 2016; 47: 9-22.
- [Background] Stickley T, Hui A, Morgan J, Bertram G. Experiences and constructions of art: a narrative-discourse analysis. J Psychiatr Ment Health Nurs. 2007 Dec;14(8):783-90. doi: 10.1111/j.1365-2850.2007.01173.x. PMID 18039303
- [Background] Davidson, L., Sells, D., Sangster, S., O'Connell, M. Qualitative studies of recovery: What can we learn from the person? In R. Ralph, & P. Corrigan (Eds.), Recovery in Mental Illness - Broadening our understanding of wellness. Washington, 2005, DC: American Psychological Association.
- [Background] Thyme, K., Sundin, E., Stahlberg, G., Lindstrom, B. Eklof, H., Wiberg, B. The outcome of short term psychodynamic art therapy compared to short term psychodynamic verbal therapy for depressed women. Psychodynamic Psychotherapy. 2007; (21): 251-264.
- [Background] Teglbjaerg HS. Art therapy may reduce psychopathology in schizophrenia by strengthening the patients' sense of self: a qualitative extended case report. Psychopathology. 2011;44(5):314-8. doi: 10.1159/000325025. Epub 2011 Jun 9. PMID 21659793
- [Background] Blomdahl, C., Gunnarsson, B., Guregard, S., Bjorklund, A. A realist review of art therapy for clients with depression. The Arts in Psychotherapy. 2013; 40(3): 322-330.
- [Background] Montag C, Haase L, Seidel D, Bayerl M, Gallinat J, Herrmann U, Dannecker K. A pilot RCT of psychodynamic group art therapy for patients in acute psychotic episodes: feasibility, impact on symptoms and mentalising capacity. PLoS One. 2014 Nov 13;9(11):e112348. doi: 10.1371/journal.pone.0112348. eCollection 2014. PMID 25393414
- [Background] Noiseux S, St-Cyr Tribble D, Leclerc C, Ricard N, Corin E, Morissette R, Lambert R. Developing a model of recovery in mental health. BMC Health Serv Res. 2009 May 1;9:73. doi: 10.1186/1472-6963-9-73. PMID 19409092
- [Result] Laranjeira C, Campos C, Bessa A, Neves G, Marques MI. Mental Health Recovery Through "Art Therapy": A Pilot Study in Portuguese Acute Inpatient Setting. Issues Ment Health Nurs. 2019 May;40(5):399-404. doi: 10.1080/01612840.2018.1563255. Epub 2019 Apr 3. PMID 30943062